CLINICAL TRIAL: NCT02836652
Title: Prevention of Non-Surgical Bleeding by Management of HeartMate II Patients Without Antiplatelet Therapy
Acronym: PREVENT II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJM-CIP-10134
Record Dates: First submitted 2016-07-12; First posted 2016-07-19 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: HeartMate II (HMII); Left Ventricular Assist Device (LVAD)
MeSH Terms: conditions — Heart Failure | interventions — Warfarin; Aspirin; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): Warfarin (INR Target 2.0-2.5, median 2.25, per standard of patient care) + placebo (1 pill/day) post HeartMate II implant
  Interventions: Device: HeartMate II (HMII); Drug: Warfarin
- Control Arm (Active Comparator): Warfarin (INR Target 2.0-2.5, median 2.25, per standard of patient care) + acetylsalicylic acid (ASA) therapy (81mg/day) post HeartMate II implant
  Interventions: Device: HeartMate II (HMII); Drug: Warfarin; Drug: acetylsalicylic acid (ASA) therapy

INTERVENTIONS:
Device: HeartMate II (HMII) — Left Ventricular Assist Device
Drug: Warfarin — (INR Target 2.0-2.5, median 2.25, per standard of patient care)
  Other Names: Coumadin
Drug: acetylsalicylic acid (ASA) therapy — (81mg/day)
  Other Names: Aspirin
  Arms: Control Arm

SUMMARY:
This study is a prospective, multi-center, randomized, double-blind placebo-controlled study of subjects receiving the HM II LVAD as per the current FDA approved indications for use.

DETAILED DESCRIPTION:
This is a post-market clinical study of HM II patient management practices to be conducted in the United States.

Subjects will be randomized in a 1:1 fashion to the following research drug groups:

1. Treatment Arm: Warfarin (INR target: 2.0-2.5, median: 2.25) + Placebo (1 pill/day)
2. Control Arm: Warfarin (INR target: 2.0-2.5, median: 2.25) + ASA Therapy (81mg/day)

The study will investigate if subjects in the Treatment Arm experience a reduced incidence of non-surgical bleeding, without an increased risk of thromboembolic events.

ELIGIBILITY:
Inclusion Criteria

* Subject is receiving the HM II per standard of care (SOC) in accordance with the FDA approved indications for use
* Subject is ≥ 50 years of age
* Subject is receiving the HM II as their first LVAD
* Subject or legally authorized representative (LAR) has signed an informed consent form (ICF).

Exclusion Criteria

* Existence of ongoing mechanical circulatory support (MCS) other than intra-aortic balloon pump or Impella® devices
* Participation in any other clinical investigation(s) involving an MCS device, or an investigation(s) that is likely to confound study results or affect study outcome
* Antiplatelet therapy is mandated for other conditions, in particular: a) recent coronary artery stenting (≤ 6 months), b) carotid artery disease, and c) other conditions where the investigator is not comfortable leaving subjects off-ASA or starting ASA post LVAD implantation. In situations where the investigator is uncertain, the Steering Committee can provide recommendation to the investigator as needed.
* Subjects in whom heart transplantation is expected in ≤ 6 months
* Subjects with a known ASA allergy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Crandall, Study Director — Abbott
Locations (35):
- United States (33):
  - University of Alabama Hospital at Birmingham (UAB), Birmingham, Alabama
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Shands at the University of Florida, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian Hospital/Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Providence St. Vincent, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Seton Medical Center, Austin, Texas
  - Baylor University Hospital, Dallas, Texas
  - Memorial Hermann, Houston, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - Institut de Cardiologie de Quebec (Hôpital Laval), Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Warfarin (INR Target 2.0-2.5, median 2.25, per standard of patient care) + placebo (1 pill/day) post HeartMate II implant
  HeartMate II (HMII): Left Ventricular Assist Device
  Warfarin: (INR Target 2.0-2.5, median 2.25, per standard of patient care)
- Aspirin: Warfarin (INR Target 2.0-2.5, median 2.25, per standard of patient care) + acetylsalicylic acid (ASA) therapy (81mg/day) post HeartMate II implant
  HeartMate II (HMII): Left Ventricular Assist Device
  Warfarin: (INR Target 2.0-2.5, median 2.25, per standard of patient care)
  acetylsalicylic acid (ASA) therapy: (81mg/day)
Period: Overall Study
Arm/Group | Placebo | Aspirin
Started | 35 | 37
As-treated Population (Cohort of subjects on treatment medication.) | 31 | 34
Completed | 17 | 18
Not Completed | 18 | 19
Not completed — Death | 3 | 3
Not completed — Transplant/Explant | 3 | 4
Not completed — Withdrawn | 9 | 9
Not completed — Not on treatment regimen post-op day 15 | 3 | 3

BASELINE CHARACTERISTICS:
Population: As-treated population: patients that consented to participate in the study and were able to start the research drug within 15 days of HM II implant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aspirin | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (5.9) | 65.6 (6.5) | 66.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 25 | 31 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 9 | 14
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72
Ischemic Heart Failure [Count of Participants; unit: Participants] | 15 | 24 | 39
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 13 | 14 | 27
History of Stroke [Count of Participants; unit: Participants] | 6 | 2 | 8
History of Bleed [Count of Participants; unit: Participants] | 1 | 5 | 6
History of Gastrointestinal Bleed [Count of Participants; unit: Participants] | 0 | 2 | 2
History of Myocardial Infarction [Count of Participants; unit: Participants] | 12 | 21 | 33
History of Diabetes [Count of Participants; unit: Participants] | 18 | 18 | 36
History of Aortic Stenosis [Count of Participants; unit: Participants] | 0 | 1 | 1
History of Carotid Artery Disease [Count of Participants; unit: Participants] | 3 | 4 | 7
Left Ventricular Ejection Fraction (%) - mean ± standard deviation (SD) [Mean (Standard Deviation); unit: %] | 18.0 (5.9) | 16.8 (5.1) | 17.4 (5.5)
Right Atrial Pressure (mm-Hg) - mean ± SD [Mean (Standard Deviation); unit: mm-Hg] | 10.5 (7.0) | 9.6 (5.5) | 10.0 (6.2)
Mean Arterial Pressure (mm-Hg) - mean ± SD [Mean (Standard Deviation); unit: mm-Hg] | 83.8 (10.3) | 85.6 (14.2) | 84.8 (12.4)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 56.2 (17.3) | 58.6 (22.0) | 57.5 (19.8)
Destination Therapy [Count of Participants; unit: Participants] — Destination therapy is when the device is implanted with the intent of having the device provide long-term or permanent support for the heart as opposed to being a bridge to heart transplant. The left ventricular assist device (LVAD) team makes this determination prior to the LVAD implant based on the patient's cardiac function and other comorbidities, which will also determine their eligibility for receiving a heart transplant.
  Participants | 28 | 29 | 57
Inter-agency Registry for Mechanically Assisted Circulatory Support (INTERMACS) <= 3 [Count of Participants; unit: Participants] — INTERMACS profiles are commonly used to identify the severity of heart failure. Simplified definitions of profiles 1-3 are listed below.
  1. The patient has life-threatening hypotension, increasing need for cardiac medications and diminishing end-organ perfusion.
  2. Progressively declining nutritional intake and renal function, fluid retention, or other major status indicator, despite being on cardiac medications.
  3. The patient is stable, has normal nutritional intake, end-organ function and is not hypotensive, but is dependent on cardiac medications.
  Participants | 28 | 26 | 54
Cardiac Re-synchronization Therapy with Defibrillator [Count of Participants; unit: Participants] | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: % of Patients With Non-surgical Bleeding at 6 Months Post HeartMate II Implant
Description: Composite incidence of non-surgical bleeding at 6 months post initial implantation, including but not limited to gastrointestinal, genitourinary, epistaxis, subdural hematoma, and primary hemorrhagic stroke (not due to ischemic conversion, or due to the treatment of a hemolysis/suspected thrombosis event).
Time Frame: 6 months post initial implantation
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 31 | 34
Participants | 12 | 15

2. Primary Outcome: Efficacy Endpoint: % of Patients With Thromboembolic Events at 6 Months Post HeartMate II Implant
Description: Composite incidence of pump thrombosis and thromboembolic stroke at 6 months post initial implantation, including ischemic stroke, or hemorrhagic stroke due to an ischemic conversion/treatment of hemolysis/pump thrombosis event.
Time Frame: 6 months post initial implantation
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 31 | 34
Participants | 4 | 3

3. Other Pre Specified Outcome: Descriptive Endpoint: Percent of Patients With Adverse Events at 1-year Post HeartMate II Implant
Description: Rates of bleeding, gastrointestinal (GI) bleeding, suspected and confirmed pump thrombosis, stroke, hemolysis, anticoagulation, survival.
Time Frame: 12 months post-implant
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 31 | 34
percentage of subjects
  Major Bleeding | 38.7 | 64.7
  GI Bleeding | 25.8 | 29.4
  Ischemic Stroke | 12.9 | 14.7
  Hemorrhagic Stroke | 6.5 | 5.9
  Transient Ischemic Attack | 9.7 | 0
  Hemolysis | 22.6 | 17.6
  Suspected Pump Thrombosis | 9.7 | 8.8
  Confirmed Pump Thrombosis | 6.5 | 5.9

4. Other Pre Specified Outcome: Adherence to Prevention of HeartMate II Pump Thrombosis Through Clinical Management (PREVENT) Study Recommended Practices
Description: The PREVENT recommended practices have three objectives: maximizing flow through the pump, reducing the risk of cannula malposition, and ensuring adequate anticoagulation while on left ventricular device support, with the overall goal of reducing pump thrombosis events. These implant techniques are similar to those in the HeartMate II instructions for use, but with modifications derived from clinical experience.
Time Frame: 12 months post-implant
Population: As-treated population
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 30 | 34
percentage of subjects
  Was the pump pocket adequately sized? | 100 | 100
  Was the pump pocket inferiorly deep and lateral? | 100 | 100
  Was the pump positioned below the diaphragm? | 100 | 100
  Was the pump anchored? | 76.7 | 85.3
  Was inflow cannula parallel to septum and oriented | 100 | 100
  Location of core: True Apex | 46.7 | 52.9
  Does the outflow graft avoid the right ventricle? | 93.3 | 100
  Was Heparin Bridging started? | 76.7 | 85.3
  Was Warfarin initiated within 48 hours post HMII i | 66.7 | 50.0
  Was a goal INR of 2.0 - 2.5 achieved in post-op da | 50.0 | 26.5
  Was the treatment drug therapy initiated within 5 | 76.7 | 73.5
  Pump speed <9000 leaving OR? | 45.2 | 41.2
  Pump speed < 9000 at 30 days? | 14.3 | 9.4

ADVERSE EVENTS:
Time Frame: At the end of study follow-up: 12-months HM II implant.
Description: Adverse events and deaths occurring in the "as-treated population" are reported here. This includes patients that consented to participate in the study and were able to start the research drug within 15 days of HM II implant.
Arm/Group | Placebo | Aspirin
All-Cause Mortality (participants affected / at risk) | 3/31 | 3/34
Serious Adverse Events (participants affected / at risk) | 21/31 | 26/34
Other Adverse Events (participants affected / at risk) | 0/31 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Aspirin (N=34)
Major Bleeding (Vascular disorders) | 12 (20) | 22 (35)
Stroke (Nervous system disorders) | 6 (6) | 7 (7)
Hemolysis (Blood and lymphatic system disorders) | 7 (7) | 6 (6)
Suspected Pump Thrombosis (Product Issues) | 3 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
1. The study did not complete enrollment due to competing enrollment in MOMENTUM 3.
2. Other adverse events were not collected in this study.
3. INR data are incomplete and hence, are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02836652/Prot_SAP_000.pdf